CLINICAL TRIAL: NCT00105898
Title: Internet-based Diabetes Education and Case Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TEL 02-100
Record Dates: First submitted 2005-03-17; First posted 2005-03-18 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2010-08

CONDITIONS: Diabetes Mellitus; Hypertension
Keywords: Diabetes mellitus; Hypertension; Telemedicine; Case management
MeSH Terms: conditions — Diabetes Mellitus; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental): Intervention group
  Interventions: Procedure: Web-based care management
- Arm 2 (Active Comparator): Comparator
  Interventions: Procedure: Telephone and face-to-face care management
- Arm 3 (Sham Comparator): Comparator
  Interventions: Procedure: Internet access alone

INTERVENTIONS:
Procedure: Web-based care management — Participants interact with a care manager, sending and receiving messages using an internet portal that accepts uploads from glucose and BP meters
  Arms: Arm 1
Procedure: Telephone and face-to-face care management — Participants interact with a care manager via face-to-face and telephone contact
  Arms: Arm 2
Procedure: Internet access alone — Participants are given internet access and encouraged to seek diabetes information to help in their self management
  Arms: Arm 3

SUMMARY:
This study is comparing the effectiveness of web-based care management to either telephone-based care management or internet access alone, in patients with poorly controlled diabetes mellitus.

DETAILED DESCRIPTION:
Background:

Patients with diabetes and elevated hemoglobin A1c (HbA1c) are at risk for diabetes-related complications. Care-management may be helpful in these patients, by providing direct contact between such high-risk patients and the healthcare system. Web-based systems have previously shown promise as a means of neutralizing access barriers such as scheduling and travel to appointments and may be of particular help in improving diabetes care.

Objectives:

We examined the efficacy of two methods of diabetes education and care management: (1) a traditional model that involved telephone contact and face-to-face encounters (2) a web-based model with access to a diabetes care management web site. We compared these interventions to a study group that received no education or care management but was provided with a computer and access to diabetes self-management websites.

Methods:

This study employed a randomized, parallel group design involving patients with diabetes mellitus and an elevated HbA1c ( 8.5%). Participants assigned to web-based care management received a notebook computer, Internet access and interacted with a care manager through a diabetes education and care management website. Participants receiving telephone-based care management interacted with a care manager using telephone and face-to-face contact. Both care management models employed medication algorithms to improve glucose and BP control. These care management groups were compared to a study group that had no care management but received a notebook computer and Internet access with their "home page" containing links to a series of diabetes self-management websites (i.e. computer only group). The primary outcome measures were HbA1c, blood pressure, and scores on the Problem Areas in Diabetes (PAID) questionnaire, each measured over 12-months.

Status:

Complete

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes mellitus
* Age 25-79 years
* HbA1c >=8.5%
* Ability to speak and understand English
* Telephone access
* VA-based primary care provider
* Interest in using a glucose and BP monitor and notebook computer

Exclusion Criteria:

* Visual impairment that affects ability to read

Ages: 25 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2005-02; Primary Completion 2007-04 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c at 12 months | 12 months

SECONDARY OUTCOMES:
Change in blood pressure, lipid profile and diabetes-related stress (self-report) at 12 months; cost-effectiveness analysis of the interventions. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul R. Conlin, MD, Principal Investigator — VA Boston Healthcare System Brockton Campus, Brockton, MA
Locations (1):
- VA Boston Healthcare System Brockton Campus, Brockton, MA, Brockton, Massachusetts, United States

REFERENCES:
- [Result] Conlin PR. Genes and environment in blood pressure control--salt intake again shows its importance. Am J Clin Nutr. 2008 Aug;88(2):255-6. doi: 10.1093/ajcn/88.2.255. No abstract available. PMID 18689358
- [Result] Kerfoot BP, Conlin PR, Travison T, McMahon GT. Patient safety knowledge and its determinants in medical trainees. J Gen Intern Med. 2007 Aug;22(8):1150-4. doi: 10.1007/s11606-007-0247-8. Epub 2007 Jun 6. PMID 17551796
- [Derived] McMahon GT, Fonda SJ, Gomes HE, Alexis G, Conlin PR. A randomized comparison of online- and telephone-based care management with internet training alone in adult patients with poorly controlled type 2 diabetes. Diabetes Technol Ther. 2012 Nov;14(11):1060-7. doi: 10.1089/dia.2012.0137. Epub 2012 Sep 6. PMID 22953754